CLINICAL TRIAL: NCT05176886
Title: Assessment of the Correct Tip Position of Central Venous Catheters, Inserted Using Patient's Height Formula
Brief Title: Correct Tip Position of Central Venous Catheters
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halide Hande Şahinkaya, MD, Anesthesiology Specialist, Bozyaka Training and Research Hospital
Other Study IDs: Catheter
Record Dates: First submitted 2021-11-27; First posted 2022-01-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Central Venous Catheter; Internal Jugular Vein; Radiography; Subclavian Vein Injury
Keywords: central venous catheter insertion; Peres' formula; correct tip position; carina

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients, ages between 18-70 years, who require central venous catheter will be enrolled for the study. Central venous catheter will be inserted using patient's height formula by Seldinger technique. Anterioposterior chest radiography will be used to assess the correct tip position. Catheters that are below the carina more than 1 cm, will be pulled back for repositioning. Catheters that are above the carina more than 1 cm, will be changed by another catheter. The investigators aim to evaluate the formula for correct tip positioning for central venous catheters

DETAILED DESCRIPTION:
Central venous catheters are used for fluid infusion, nutrition, blood transfusion, hemodynamic monitorization in both intensive care unit and operating room. The superior vena cava and right atrium (SVC-RA) junction is considered the optimal position for central venous catheter tip. Carina corresponds to the SVC-RA junction on chest radiograph. Catheter tips, 1 cm above and 1 cm below the carina are considered as the correct position. 18-70 years old patients will be enrolled for the study. Central venous catheters will be inserted via internal jugular vein or subclavian vein using patient's height formula by Seldinger technique. Postprocedural (within 6 hours) chest radiograph will be used to evaluate the correct tip position from the Picture Archiving and Communication System. This formula was described by Peres. If the tip of the catheter is below the carina more than 1 cm, it will be pulled back for repositioning. If the tip of the catheter is above the carina more than 1 cm, another catheter will be inserted. The formula is height (cm)/10 for right internal jugular vein, height(cm)/10-2 for right subclavian vein, height(cm)/10+4 for left internal jugular vein and height(cm)/10+2 for left subclavian vein. Number of the correct and incorrect position of central venous catheter tips will be noted.

The investigators aim to evaluate the reliability and efficiency of Peres' formula for the correct tip position.

ELIGIBILITY:
Inclusion Criteria:

* Central venous catheterization of patients, ages between 18 and 70

Exclusion Criteria:

* Patient's refusal
* Pathology of carotid artery
* Anatomical deformity of the neck (scar, mass effect, multiple central venous catheterization)
* Chest deformities (pectus excavatum, pectus carinatum)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care unit and operating room who require a central venous catheter (right or left-sided) will be enrolled for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of correct position of central venous catheter tip | Within 6 hours after placement of central venous catheter
  Central venous catheter tip should be placed at the superior vena cava and right atrium junction. This junction is defined as carina in anteroposterior chest x-ray imagining. Correct tip position is defined as 1 cm above and 1 cm below the carina.Postprocedural chest radiography will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Halide H Şahinkaya, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Mine Parlak, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Zeki T Tekgül, MD, Study Chair — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi AM, Bhosale GP, Parikh GP, Shah VR. Optimal positioning of right-sided internal jugular venous catheters: comparison of intra-atrial electrocardiography versus Peres' formula. Indian J Crit Care Med. 2008 Jan;12(1):10-4. doi: 10.4103/0972-5229.40943. PMID 19826584
- [Background] Kujur R, Rao MS, Mrinal M. How correct is the correct length for central venous catheter insertion. Indian J Crit Care Med. 2009 Jul-Sep;13(3):159-62. doi: 10.4103/0972-5229.58543. PMID 20040815
- [Background] Salimi F, Imani MR, Ghasemi N, Keshavarzian A, Jazi AH. The mid-sternal length, a practical anatomical landmark for optimal positioning of long-term central venous catheters. J Res Med Sci. 2013 May;18(5):383-6. PMID 24174941